CLINICAL TRIAL: NCT04735640
Title: Effects of a 9-months Nurse-led Telephone Personalized Lifestyle Intervention Versus Automated SMSs on Nutritional and Physical Activity Advice on Glucose Profile in Patients With Prediabetes
Brief Title: Effectiveness of a Nurse-led Personalized Telephone Intervention on Lifestyle Changes in Diabetes Prevention.
Acronym: PREDIPHONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Josep1, PhD, University of the Balearic Islands
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI18/01209
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Prediabetic State
Keywords: prediabetes; type 2 diabetes; fasting plasma glucose; diet; physical activity; randomized clinical trial
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-led teleconsultation group (Experimental): 9-month nurse-led telephone-based personalized behavioural intervention.
  Interventions: Behavioral: nurse-led teleconsultation
- SMS group (Active Comparator): Behavioural intervention by means of short text messages.
  Interventions: Behavioral: SMS

INTERVENTIONS:
Behavioral: nurse-led teleconsultation — Patients assigned to this group will receive personalized dietary and physical activity advice during 9 months. Behavioural goals and action plans will be developed in a stepwise manner in accordance with baseline levels of nutritional and physical activity adherence to recommendations.
  Arms: Nurse-led teleconsultation group
Behavioral: SMS — Patients assigned to this group will receive a total of 150 text messages (4 to 5 messages per week during weekdays) throughout the intervention period (9 months). The content of the text messages includes advice on diet and exercise.
  Arms: SMS group

SUMMARY:
A randomized, 9-months, parallel-group study comparing the effectiveness of a nurse-led telephone personalized lifestyle intervention versus automated SMSs on nutritional and physical activity advice in the reduction of fasting blood glucose and/or HbA1c in a population with prediabetes.

DETAILED DESCRIPTION:
It is estimated that about 70% of the prediabetic population will eventually develop type 2 diabetes (T2DM), contributing to the significant economic burden on health systems and societies. When prediabetes is recognized, lifestyle intervention including weight loss through diet and exercise can reduce the relative risk of developing T2DM by more than 50% within 3 years. In the context of the current pandemic caused by COVID-19 the implementation of prevention strategies is heavily affected. Telemedicine consultations give patients the opportunity to receive personalized advice on disease prevention even in times of pandemic. Previous studies on telemedicine intervention strategies for the prevention of T2DM show that there is a need to further explore the utility of telemedicine and especially telephone-based personalized behavioural interventions in patients with prediabetes.The aim of the present research is to determine whether a nurse-led personalized telephone lifestyle intervention is effective in reducing risk factors associated with the development of T2DM in subjects with prediabetes, versus automated short message service (SMS).

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma glucose between 100 and 125 mg/dL OR HbA1c between 5.7 and 6.4%
* BMI ≥ 27 and < 40 kg/m2
* Written informed consent

Exclusion Criteria:

* Documented history of T2DM or use of oral antidiabetic medication
* Terminal illness
* Institutionalization, dementia or cognitive impairment
* Pregnancy
* Major surgery or hospital stay during the previous 3 months
* Documented history of hematologic disease which may interfere with the HbA1c measurement
* Presence of any medical or psychological condition that may limit the ability of the patient to participate in the study
* Concomitant active participation in another clinical trial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Change in fasting plasma glucose | at baseline, 4, 9, and 15 months
  Change in fasting plasma glucose at 4, 9, and 15 months versus baseline

SECONDARY OUTCOMES:
Blood levels of HbA1c | at baseline, 4, 9, and 15 months
  Change in HbA1c levels at 4, 9, and 15 months versus baseline
Maintenance of acquired dietary and physical activity changes | 15 month
  Whether lifestyle changes acquired during the 9-month active-intervention phase are maintained in the mid-term.

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Bennasar Veny, PhD, Principal Investigator — University of the Balearic Islands
Locations (1):
- University of the Balearic Islands, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arias-Fernandez M, Huguet-Torres A, Abbate M, Fresneda S, Torres-Carballo M, Carvalho-Azevedo A, Yanez AM, Bennasar-Veny M. Effectiveness of a low-intensity nurse-led lifestyle intervention on glycaemic control in individuals with prediabetes: The PREDIPHONE randomized controlled clinical trial. Int J Nurs Stud. 2025 May;165:105034. doi: 10.1016/j.ijnurstu.2025.105034. Epub 2025 Feb 22. PMID 40058011
- [Derived] Abbate M, Fresneda S, Yanez A, Ricci-Cabello I, Galmes-Panades AM, Aguilo A, Bennasar-Veny M; PREDIPHONE trial group. Nurse-led telephone intervention for lifestyle changes on glycaemic control in people with prediabetes: Study protocol for a randomized controlled trial. J Adv Nurs. 2021 Jul;77(7):3204-3217. doi: 10.1111/jan.14842. Epub 2021 Mar 26. PMID 33769603